CLINICAL TRIAL: NCT02281513
Title: Activity and Nutrition Trial in Lupus to Energize and Renew
Acronym: ANTLER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Rosalind Ramsey-Goldman, Solovy Arthritis Research Society Research Professor of Medicine, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STU 69201
Record Dates: First submitted 2014-10-22; First posted 2014-11-03 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Systemic Lupus Erythematosus; Physical Activity; Sleep
Keywords: Nutrition
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Motor Activity | interventions — pilose antler peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ANTLER Pilot Cohort (Other): Pilot study participants will be provided the smartphone application, fitbit activity monitor, and coaching sessions.
  Interventions: Other: Smartphone Application; Other: Fitbit Activity Monitor; Other: Coaching Sessions

INTERVENTIONS:
Other: Smartphone Application — Is a self-monitoring tool to document fruit and vegetable consumption, sleep quantity and quality, and physical activity
  Other Names: ANTLER
Other: Fitbit Activity Monitor — Is connected to this smartphone application so that participants who wear this monitor have data that automatically populates the smartphone application for physical activity.
Other: Coaching Sessions — Using motivational interviewing (a counseling style used in helping persons change their behavior) at baseline after completion of all baseline assessments and at follow up after completion of all follow up assessments. Coaching session includes discussion of facilitators and barriers to increasing physical activity, fruit and vegetable consumption and sleep, as well as setting goals to work towards at next meeting. The coach will monitor the information that the participant enters into the smartphone application and will provide feedback on a weekly basis to the participant.

SUMMARY:
Participants from the Fatigue and Lifestyle Physical Activity and SLE Study will be approached to enroll in a 6 week pilot intervention. This study will look at the barriers and facilitators to increasing physical activity, improving dietary/nutritional intake, and improving sleep.This study will offer support and information for people with SLE to increase their physical activity, improve their dietary/nutritional intake, and improve their sleep and will utilize a smartphone application to self-monitor changes in these behaviors.

DETAILED DESCRIPTION:
Description of ANTLER pilot intervention: a 6 week intensive program which combines the following goals

* Ability of participants to utilize a smart phone application for self-monitoring behavior change of physical activity, fruit/vegetable consumption, and sleep. This would include entering data on fruit/vegetable consumption, hours of sleep and monitoring feedback.
* Ability of participants to wear Actigraph accelerometer 24 hours/day and complete a sleep log for measurement of physical activity and sleep.
* Ability of Nutrition Data System for Research (NDSR) software to collect adequate nutrition data.

The intervention is a unique combination of two individual counseling sessions and the utilization of a combination of a smartphone application and the use of a Fitbit physical activity monitor. The individual sessions will provide a tailored personalized intervention including problem-solving and goal setting for increasing physical activity, consumption of more fruits and vegetables, and getting more sleep. Healthy Lifestyle Coaches (RN or Exercise Physiologist) will be responsible for conducting the individual sessions for a limited caseload of participants.

Individual sessions will

* utilize motivational interviewing techniques to enhance motivation for meeting individualized physical activity, dietary/nutritional and sleep goals
* identify specific barriers and supports leading to tailored intervention to increase program success (The Arthritis Comprehensive Treatment Assessment)
* provide emotional support

Self-monitoring of behavior change

* On a daily basis, participants will log fruit/vegetable consumption and hours of sleep via a smartphone application and receive feedback
* On a daily basis, participants will monitor their physical activity via the Fitbit and receive feedback on the smartphone.

Online activities will include communication between the client and coach in between and after scheduled intervention visits.

ELIGIBILITY:
Inclusion Criteria:

* 1) meet at least 4 of 11 ACR classification criteria for definite SLE 2) at least 18 years of age, 3) BMI between 14 and 40 kg/m2, 4) able to ambulate at least household distances (50ft), 5) ability to complete the dietary recall assessment, and 6) able to provide informed consent.

After informed consent is obtained, a medical record review will determine whether there is a history of uncontrolled diabetes mellitus or cardiovascular disease. Potential participants will be asked to complete the PAR-Q to determine restriction in physical activity. Blood pressure will be assessed and potential participants will be excluded if SBP>160 or DBP >110.

Exclusion Criteria:

* Does not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Measurement of Fatigue | Up to 6 weeks
  It is measured by the Fatigue Severity Scale and the PROMIS Fatigue Short-Form online via the Assessment Center. Change from baseline to 6-week follow-up is measured. The Fatigue Severity Scale is 9 items scored on a 7-point scale from 1= strongly disagree to 7=strongly agree. Minimum score =9 and maximum score=63. Higher score=greater fatigue severity. The PROMIS Fatigue Short Form is 8 items looking back at the past 7 days assessing amount of fatigue and trouble getting things done because of fatigue on a 5-point scale.

SECONDARY OUTCOMES:
PA, Diet Assessments and Sleep | Up to 6 weeks
  Physical activity is measured objectively by accelerometer worn for 7 days, 24 hours per day and maintenance of a sleep log and self-report of activity by the International Physical Activity Questionnaire (IPAQ) by interview based on the 7 days that the accelerometer is worn. Fruit/vegetable consumption is measured by the Nutrition Data System for Research per interview. Sleep is measured by the PROMIS sleep disturbance and sleep-related impairment Short Forms online via the Assessment Center. Change from baseline to 6-week follow-up is measured for all of these secondary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind Ramsey-Goldman, MD, DrPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Plans for Resource Sharing. The final data sets from this project will include lupus disease and damage measurements, raw and processed nutrient intake, raw and processed patient-reported outcomes, raw and processed accelerometer data, and motivational interviewing data. The final data from this project will be de-identified in accordance with HIPAA guidelines. Prior to any type of sharing, all disease activity, nutrient intake, patient-reported outcomes and accelerometer records will be made anonymous by the assignment of a new, unique subject identifier that is not linked to any clinical medical record. Requests for resource sharing will all meet the necessary IRB requirements from Northwestern University and the institution of the individual who requests the data.

REFERENCES:
- [Background] Mancuso CA, Perna M, Sargent AB, Salmon JE. Perceptions and measurements of physical activity in patients with systemic lupus erythematosus. Lupus. 2011 Mar;20(3):231-42. doi: 10.1177/0961203310383737. Epub 2010 Dec 23. PMID 21183562
- [Background] Chandrasekhara PK, Jayachandran NV, Rajasekhar L, Thomas J, Narsimulu G. The prevalence and associations of sleep disturbances in patients with systemic lupus erythematosus. Mod Rheumatol. 2009;19(4):407-15. doi: 10.1007/s10165-009-0185-x. Epub 2009 Jun 12. PMID 19521744
- [Background] Da Costa D, Bernatsky S, Dritsa M, Clarke AE, Dasgupta K, Keshani A, Pineau C. Determinants of sleep quality in women with systemic lupus erythematosus. Arthritis Rheum. 2005 Apr 15;53(2):272-8. doi: 10.1002/art.21069. PMID 15818653
- [Background] Ehrlich-Jones L, Mallinson T, Fischer H, Bateman J, Semanik PA, Spring B, Ruderman E, Chang RW. Increasing physical activity in patients with arthritis: a tailored health promotion program. Chronic Illn. 2010 Dec;6(4):272-81. doi: 10.1177/1742395309351243. Epub 2010 Aug 9. PMID 20696695
- [Background] Stephens J, Allen J. Mobile phone interventions to increase physical activity and reduce weight: a systematic review. J Cardiovasc Nurs. 2013 Jul-Aug;28(4):320-9. doi: 10.1097/JCN.0b013e318250a3e7. PMID 22635061
- [Background] Miller W, Rollnick S. Motivational Interviewing: Preparing People for Change. 2nd edition ed. New York: Guilford Press; 2002.
- [Background] Burke LE, Wang J, Sevick MA. Self-monitoring in weight loss: a systematic review of the literature. J Am Diet Assoc. 2011 Jan;111(1):92-102. doi: 10.1016/j.jada.2010.10.008. PMID 21185970
- [Background] Hutchesson MJ, Rollo ME, Callister R, Collins CE. Self-monitoring of dietary intake by young women: online food records completed on computer or smartphone are as accurate as paper-based food records but more acceptable. J Acad Nutr Diet. 2015 Jan;115(1):87-94. doi: 10.1016/j.jand.2014.07.036. Epub 2014 Sep 26. PMID 25262244
- [Background] Mohr DC, Cuijpers P, Lehman K. Supportive accountability: a model for providing human support to enhance adherence to eHealth interventions. J Med Internet Res. 2011 Mar 10;13(1):e30. doi: 10.2196/jmir.1602. PMID 21393123
- [Background] Matthews CE, Ainsworth BE, Thompson RW, Bassett DR Jr. Sources of variance in daily physical activity levels as measured by an accelerometer. Med Sci Sports Exerc. 2002 Aug;34(8):1376-81. doi: 10.1097/00005768-200208000-00021. PMID 12165695
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] Warburton DE, Gledhill N, Jamnik VK, Bredin SS, McKenzie DC, Stone J, Charlesworth S, Shephard RJ. Evidence-based risk assessment and recommendations for physical activity clearance: Consensus Document 2011. Appl Physiol Nutr Metab. 2011 Jul;36 Suppl 1:S266-98. doi: 10.1139/h11-062. PMID 21800945
- See also: Lupus Research Program Website — http://lupus.northwestern.edu/index.html